CLINICAL TRIAL: NCT02138474
Title: The Efficacy of Lacticum Acidum Homaccord in the Treatment of Chronic Tension-type Headaches
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Johannesburg (Other)
Responsible Party: Principal Investigator, Dr J. Pellow, Dr, University of Johannesburg
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Maimela200904978; Maimela (Other: HDC43/02-2010)
Record Dates: First submitted 2014-05-12; First posted 2014-05-14 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Chronic Tension-type Headaches
Keywords: Lacticum acidum homaccord; homeopathy; chronic tension-type headaches

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lacticum acidum homaccord (Experimental): Lacticum acidum homaccord 30 mL bottle of medicated sucrose pillules take 5 pillules of the medication in the morning and in the evening for 4 weeks
  Interventions: Other: Lacticum acidum homaccord
- Placebo (Placebo Comparator): Unmedicated sucrose pillules, take 5 pillules twice daily for 4 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Lacticum acidum homaccord — Homeopathic remedy, made using sucrose pillules
  Arms: Lacticum acidum homaccord
Other: Placebo — Unmedicated sucrose pillules
  Arms: Placebo

SUMMARY:
Chronic tension-type headaches (CTTHs) affect 30-40% of the population and account for a number of absences from, and decreased performances at, work and school as well as recreational activities. CTTHs typically occur at least 15 times a month or at least every second day, and present as an achy or tight sensation that is felt around the head . The pain may last from 30 minutes to several days and varies in intensity . Conventional treatment is palliative, consisting of analgesics and non-steroidal anti-inflammatory drugs (NSAIDs), which may produce adverse effects and analgesic rebound headaches . Lacticum acidum 30CH is a homoeopathic remedy that has been shown to have potential benefits in the treatment of CTTHs . Homaccords are the preparation of one remedy in multiple increasing potencies in a single vehicle . There has been no research done to date on Lacticum acidum Homaccord in the treatment of CTTHs.The aim of this study is to determine the efficacy of Lacticum acidum Homaccord in the treatment of chronic tension-type headaches, using the modified Headache Diary and the Headache Disability Inventory.

DETAILED DESCRIPTION:
The study will be a four-week, double-blind, placebo-controlled study which will take place at the Homoeopathic Health Centre at the University of Johannesburg (UJ) Doornfontein campus. A randomized sample of 30 male and female participants between the ages of 18 and 45 years who suffer from CTTHs will be recruited. This will be done by means of purposive sampling via advertisements placed on the UJ campuses, with relevant permission given . At the initial consultation (day 0), prospective participants will be requested to sign the Participant Information and Consent Form . They will then complete the Screening Questionnaire to assess their eligibility for participating in the study. Those participants who meet the diagnostic criteria for CTTHs, and whose symptoms match at least eight out of the twelve Lacticum acidum headache related symptoms, will be eligible to participate. All participants will also be requested to complete a Headache Disability Inventory. Participants will be placed into matched pairs according to age and gender and will receive one 30 mL bottle of their medication. On days 1-28 each participant will be requested to complete the Headache Diary at the end of each day and to take 5 pillules of the medication in the morning and in the evening. The first follow-up visit will occur on day 14; here participants will complete the Headache Disability Inventory, the completed headache diaries will be exchanged with new ones, a relevant physical examination including vital signs will be conducted and an additional bottle of medication will be given. The final follow-up visit will occur on day 28, where each participant will complete the Headache Disability Inventory, and a relevant physical examination including vital signs will be recorded.

Collected data will be evaluated using frequencies, descriptive tests and cross tabulation, the Shapiro Wilk test, the Independent samples t-test or Mann-Whitney test, and the Friedman and Wilcoxon signed ranks tests. A possible outcome is that Lacticum acidum may have an ameliorating effect on CTTHs and may provide a possible alternative treatment option for this condition, opening up the field for further research.

ELIGIBILITY:
Inclusion Criteria:

* Are male or female participants between the ages of 18 and 45 years;
* Fit the diagnostic criteria for CTTHs: headache occurring for 15 days a month or more, for a period of more than 3 months a year and lasts for hours or may be continuous. The headache should have at least one of the following characteristics: 1. bilateral location; 2. pressing/tightening (non-pulsating) quality; 3. mild or moderate intensity, 4. aggravated by normal physical activities such as walking or climbing stairs; and at least one of the characteristics in the following categories: 5.1. photophobia, phonophobia or mild nausea, and 5.2. moderate or severe nausea or vomiting ; and
* Fit eight out of the twelve headache-related symptom criteria for Lacticum acidum .

Exclusion Criteria:

* Have history of headache or a change in their normal pattern or type of headache over the previous three months;
* Have had any head, neck or back injury in the previous month;
* Suffer from rheumatoid arthritis, a suspected tumour or vision problems;
* Use opioids or analgesics for more than 15 days a month, for more than three months a year;
* Use chronic medication such as corticosteroids, antidepressants, anti-hypertensives; and / or
* Are pregnant or breastfeeding.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-04; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
modified Headache Diary and the Headache Disability Inventory. | one month

CONTACTS AND LOCATIONS:
Overall Officials: Radmila Razlog, M.Tech Hom, Study Chair — UJ
Locations (1):
- UJ, Johannesburg, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: No